CLINICAL TRIAL: NCT01265303
Title: OPTIMIZING DIAGNOSTICS AND THERAPY OF ARRHYTHMIA AND SYNCOPE EVENTS USING INTELLIGENT TELEMETRIC SOLUTIONS - Evaluation of Arrhythmia Treatment Efficacy
Brief Title: Telemetric Arrhythmia and Syncope Diagnosis - Evaluation of Arrhythmia Treatment Efficacy
Acronym: TELEMARC 4
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Institute of Cardiology, Warsaw, Poland (Other)
Responsible Party: Prof Lukasz Szumowski, Institute of Cardiology, Warsaw Poland
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: UDAPOIG.01.03.01-00-068/09-00D
Record Dates: First submitted 2010-12-22; First posted 2010-12-23 (Estimated); Last update posted 2013-05-07 (Estimated); Status verified 2013-05

CONDITIONS: Atrial Fibrillation; Arrhythmias, Cardiac
Keywords: ablation, cardiac arrhythmia, atrial fibrillation, telemonitoring, telemetry
MeSH Terms: conditions — Atrial Fibrillation; Arrhythmias, Cardiac

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Catheter ablation (Other)
  Interventions: Device: Prolonged telemetric Full Disclosure ECG recording.
- Pacemaker implantation (Other)
  Interventions: Device: Prolonged telemetric Full Disclosure ECG recording.
- Pharmacotherapy (Other)
  Interventions: Device: Prolonged telemetric Full Disclosure ECG recording.

INTERVENTIONS:
Device: Prolonged telemetric Full Disclosure ECG recording. — Continuous Full Disclosure Telemetric ECG monitoring lasting 14 days
  Other Names: Medicalgorithmics, PocketECG

SUMMARY:
The purpose of this study is to assess efficacy of prolonged Full Disclosure ECG monitoring and signal analysis using advanced GSM telemetric technology to prescribe the most appropriate treatment of arrhythmia.

DETAILED DESCRIPTION:
Non-invasive methods enabling long-term ECG monitoring in patients with paroxysmal symptoms, such as tachycardia or palpitations increase the probability of detecting infrequent but dangerous events with profound clinical significance. Patients with recommendation for the first catheter ablation of Paroxysmal Atrial Fibrillation in the reference center will be included in the study. Eligible patients will have 14-day telemetric ECG monitoring. Based on detected arrhythmia events, patient's medical history and available documentation the most appropriate treatment will be recommended. Patients will undergo invasive procedures of ablation or pacemaker implantation or can be treated pharmacologically. After the invasive treatment or initiation of pharmacotherapy the 14-day telemetric ECG monitoring will be repeated to assess efficacy of the treatment.

Patients with no record of arrhythmia requiring treatment during the first 14 days ECG monitoring will terminate participation in the study. The referring physician will be informed. Further diagnosis or treatment should be performed at the referring physician's center according to the best clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Age - between 18 and 80 years old
* Physician recommendation for ablation treatment of arrhythmia
* Patient informed consent
* Declarative and feasible compliance (patient understands basic instructions regarding device use)

Exclusion Criteria:

* Inability to comply with the study protocol
* Lack of patient cooperation

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360 (Estimated)
Dates: Start 2011-02; Primary Completion 2014-03 (Estimated); Study Completion 2014-03 (Estimated)

PRIMARY OUTCOMES:
Occurence of atrial fibrillation | 14 days since the start of monitoring
  Confirmation of indication for catheter ablation of atrial fibrillation by detection of incidence of AF event during 14 days ECG monitoring

SECONDARY OUTCOMES:
Therapy efficacy analysis | 14 days
  The mean atrial fibrillation burden reduction
Indication for treatment other than catheter ablation | 14 days
  Confirmation of indication for treatment other than catheter ablation such as: pacemaker or pharmacotherapy by detetion of:
  1. arrhythmia other than AF qualifying for treatment
  2. Bradycardia < 40 BPM
  3. Pauses > 2,5 s on sinus rhythm or > 3,5 on AF
Correlation of patient self assessment based on the Quality of Life questionnaire and European Heart Rhythm Association (EHRA) scale with cardiac arrhythmia occurrence. | 14 days
Evaluation of stroke and bleeding risk factors incidence based on scores proposed in the European Society of Cardiology (ESC) guidelines: CHADS2VASC2 and HAS-BLED | 14 days

CONTACTS AND LOCATIONS:
Overall Officials: Lukasz J Szumowski, MD, PhD, Study Chair — National Institute of Cardiology, Warsaw, Poland
Locations (3):
- Universitair Ziekenhuis Brussel Centre for Heart- and Vascular diseases, Brussels, Belgium
- Poland (2):
  - Klinika Kardiologii CMKP, Warsaw
  - Institute of Cardiology, Warsaw